CLINICAL TRIAL: NCT06862791
Title: A Phase IIb Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of Co-administration of AZD9550 and AZD6234 in Participants Living With Obesity or Overweight With Co-morbidity (ASCEND)
Brief Title: A Weight Loss Study Evaluating Subcutaneous Treatment With AZD9550 and AZD6234 in Combination Against Placebo or Each of the Drugs Alone
Acronym: ASCEND
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8460C00004; 2024-516176-15-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2025-02-14; First posted 2025-03-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obesity or Overweight
Keywords: Obesity; Overweight; AZD9550; AZD6234
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Arm 1 (Experimental): AZD9550 low dose + AZD6234 low dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 2 (Experimental): AZD9550 medium dose + AZD6234 medium dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 3 (Experimental): AZD9550 high dose + AZD6234 high dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 4 (Experimental): AZD9550 low dose + AZD6234 medium dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 5 (Experimental): AZD9550 medium dose + AZD6234 low dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 6 (Experimental): AZD9550 high dose + AZD6234 medium dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 7 (Experimental): AZD9550 medium dose + AZD6234 high dose or placebos
  Interventions: Drug: AZD9550; Drug: AZD6234; Drug: Placebo comparator
- Arm 8 (Experimental): AZD9550 high dose or placebo
  Interventions: Drug: AZD9550; Drug: Placebo comparator
- Arm 9 (Experimental): AZD6234 high dose or placebo
  Interventions: Drug: AZD6234; Drug: Placebo comparator

INTERVENTIONS:
Drug: AZD9550 — IMP injected subcutaneous, once weekly. Unit dose strength as per CSP
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Arm 6; Arm 7; Arm 8
Drug: AZD6234 — IMP injected subcutaneous, once weekly. Unit dose strength as per CSP.
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Arm 6; Arm 7; Arm 9
Drug: Placebo comparator — Placebo matching IMP dose injected subcutaneously, once weekly.

SUMMARY:
The purpose of this study is to determine whether treatment with AZD9550 when given in combination with AZD6234 as once weekly subcutaneous (SC) injections is superior to placebo or either agent administered as monotherapy for weight loss in participants living with obesity or overweight with at least one weight-related co-morbidity.

DETAILED DESCRIPTION:
This is a Phase IIb, global, randomised, parallel-group, double-blind, placebo-controlled, multi-centre, reduced factorial study designed to evaluate the efficacy, safety and tolerability of treatment with AZD9550 and AZD6234 in combination or as monotherapy in adults who are living with obesity or overweight with at least one of the following weight-related co-morbidities: hypertension, dyslipidemia or obstructive sleep apnoea. The study is composed of a screening period, a treatment period and a follow up period with participants expected to be in the study for approximately 47 weeks. The study will be conducted at around 60 sites and in approximately 7 countries with about, 360 participants will be randomly assigned to study intervention or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 75 years of age inclusive.
* BMI: ≥ 30 kg/m2, or ≥ 27 kg/m2 with at least one weight related comorbidity.
* A stable, self-reported body weight for 3 months prior to screening.
* Male and female participants: Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participants must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History of any clinically important disease or disorder, which, in the opinion of the Investigator, may put the participant at risk.
* History or presence of GI, renal, hepatic disease.
* Previous or planned bariatric surgery or fitting of a weight loss device.
* Obesity induced by endocrine disorders such as Cushing's syndrome, insulinoma or Prader-Willi syndrome.
* History of T1DM or T2DM or symptoms indicative of insulinopenia or poor glucose control.
* HbA1c ≥ 6.5% (48 mmol/mol), fasting serum glucose ≥ 126 mg/dL (7.0 mmol/L) or random glucose ≥ 200 mg/dL (11.1 mmol/L).
* Significant gastric and hepatobiliary disease.
* History of acute or chronic pancreatitis or pancreatic amylase or lipase > 2 × ULN at screening.
* History of psychosis or bipolar disorder.
* History of major depressive disorder within the 2 years prior to screening or depression.
* Treatment with a GLP1 containing preparation, either as part of treatment or while participating in another clinical study within the 3 months or 5 half-lives of the drug prior to screening.
* Vulnerable populations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight from baseline after 36 weeks of treatment | 36 weeks
  To determine whether treatment with AZD9550 and AZD6234 in combination is superior to placebo for weight loss
Weight loss ≥ 5% from baseline after 36 weeks of treatment | 36 weeks
  To assess the effect of treatment with AZD9550 and AZD6234 in combination vs placebo on the proportion of participants with weight loss ≥ 5%

SECONDARY OUTCOMES:
Absolute change in body weight from baseline after 36 weeks of treatment | 36 weeks
  To determine whether treatment with AZD9550 and AZD6234 in combination is superior to placebo for weight loss
Absolute change in body weight from baseline after 36 weeks of treatment | 36 weeks
  To determine whether treatment with AZD9550 and AZD6234 in combination is superior to AZD9550 and AZD6234 monotherapy, and whether AZD9550 and AZD6234 as monotherapies are superior to placebo for weight loss
Weight loss ≥ 5% from baseline after 36 weeks of treatment | 36 weeks
  To assess the effect of treatment with AZD9550 and AZD6234 in combination vs monotherapy, and assess the effect of AZD9550 and AZD6234 as monotherapies vs placebo, on the proportion of participants with weight loss ≥ 5%
Weight loss ≥ 10% and ≥ 15% from baseline after 36 weeks of treatment | 36 weeks
  To assess the effect of treatment with AZD9550 and AZD6234 in combination vs placebo and monotherapy, and assess the effect of AZD9550 and AZD6234 as monotherapies vs placebo, on the proportion of participants with weight loss ≥ 10% and ≥ 15%
Prevalence of ADAs to AZD9550 and AZD6234 in combination and as monotherapies after 36 weeks of treatment | 36 weeks
  To assess the immunogenicity profile of treatment with AZD9550 and AZD6234 in combination and as monotherapies
Incidence of ADAs to AZD9550 and AZD6234 in combination and as monotherapies after 36 weeks of treatment | 36 weeks
  To assess immunogenicity profile of ADAs to AZD9550 and AZD6234 in combination and as monotherapies
Titres of ADAs to AZD9550 and AZD6234 in combination and as monotherapies after 36 weeks of treatment | 36 weeks
  To assess the immunogenicity profile of treatment with AZD9550 and AZD6234 in combination and as monotherapies
Percent change in body weight from baseline after 36 weeks of treatment | 36 weeks
  To determine whether treatment with AZD9550 and AZD6234 in combination is superior to AZD9550 and AZD6234 monotherapy, and whether AZD9550 and AZD6234 as monotherapies are superior to placebo for weight loss

CONTACTS AND LOCATIONS:
Locations (51):
- United States (29):
  - Research Site, Dothan, Alabama
  - Research Site, Vestavia Hills, Alabama
  - Research Site, Cerritos, California
  - Research Site, Escondido, California
  - Research Site, Huntington Park, California
  - Research Site, Lincoln, California
  - Research Site, Sacramento, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Palm Harbor, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, South Bend, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Sioux City, Iowa
  - Research Site, Southfield, Michigan
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Albuquerque, New Mexico
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Kingsport, Tennessee
  - Research Site, Brownsville, Texas
  - Research Site, Houston, Texas
  - Research Site, Arlington, Virginia
  - Research Site, Renton, Washington
- Australia (5):
  - Research Site, Maroochydore
  - Research Site, Maroubra
  - Research Site, Norwood
  - Research Site, St Albans
  - Research Site, St Leonards
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Montreal, Quebec
- Germany (6):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Falkensee
  - Research Site, Hamburg
  - Research Site, Münster
  - Research Site, Oldenburg
- Japan (4):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: 20260129-draft-structured-data-ascend-sm-04-de — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8460C00004&attachmentIdentifier=d1c763ba-d73e-4d0c-b946-68522269d77f&fileName=20260129-draft-structured-data-ascend-sm-04-de.pdf&versionIdentifier=